CLINICAL TRIAL: NCT02208687
Title: Energetic, a Self Management Group Program Aimed at Reconditioning and Social Participation in Persons With a Muscle Disease; a Multicentre Randomized Controlled Trial.
Brief Title: Effectiveness and Cost-effectiveness of the Energetic Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Revalidatiefonds Nederland (Unknown); Center of expertise Sneller herstel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/077
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2016-04

CONDITIONS: Neuromuscular Diseases
Keywords: Social Participation; Fatigue; Self-Management; Rehabilitation; Physical therapy; Occupational therapy; Group intervention; Exercise
MeSH Terms: conditions — Neuromuscular Diseases; Fatigue; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energetic (Experimental): Self management group program aimed at reconditioning and social participation
  Interventions: Behavioral: Energetic
- Control group (Other): Usual care
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Energetic — Physiotherapy and occupational therapy aimed at reconditioning and social participation.
  Arms: Energetic
Other: Control group — Usual care
  Arms: Control group

SUMMARY:
Fatigue is present in at least 60% of the patients with a muscle disease and can be the most disabling symptom. In combination with other impairments, this often results in low levels of physical activity and decreased social participation, leading to large societal costs. Energetic is a self-management group program aimed at improving participation and physical endurance in these patients. Our hypothesis is that Energetic results in improved participation and improved physical endurance, less experienced fatigue and better quality of life compared to usual care, without increasing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* formal diagnosis of muscular disease, either FascioScapuloHumeral Dystrophy (FSHD), Inclusion Body Myositis (IBM), Mitochondrial Myopathy (MM) or any other;
* being severely fatigued
* being cardiopulmonary stable and capable of aerobic training (as determined using a submaximal cycling exercise test with ECG (electrocardiography) and advice from a consultant cardiologist and pulmonologist);
* being motivated, committed to the program, and 'ready to change' which is discussed with the patient during the screening by a rehabilitation physician and an occupational therapist; to this end, motivational interviewing will be used (including a advantages/disadvantages matrix; a visual analogue scale (VAS) to rate the importance of participation in de program; and a VAS to rate the confidence a patient has that participation in the program is feasible)
* being able to formulate at least 3 individual participation goals during the interview with the occupational therapist.

Exclusion Criteria:

* active depression or other psychiatric disorder as indicated by a consultant psychologist or by the medical history,
* pregnancy,
* severe co-morbid condition,
* having participated in the Energetic program before
* a travel distance perceived as too burdensome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 3 months
  Perceived activity performance. Three months will be the primary analysis. Effects at follow up will be measured at 6 and 12 months (see secondary outcome measures) (patient)

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM-satisfaction) | 3 months
  Perceived satisfaction with performance (patient)
Canadian Occupational Performance Measure (COPM-satisfaction) | 6 months
  Perceived satisfaction with performance (patient)
Canadian Occupational Performance Measure (COPM-satisfaction) | 15 months
  Perceived satisfaction with performance (patient)
Canadian Occupational Performance Measure (COPM-performance) | 6 months
  Perceived performance in activities. Is primary outcome measure at 3 months, but data of 6 and 15 months follow up wil be used in a secondary analysis. (patient)
Canadian Occupational Performance Measure (COPM-performance) | 15 months
  Perceived performance in activities. Is primary outcome measure at 3 months, but data of 6 and 15 months follow up wil be used in a secondary analysis. (patient)
Activity Card Sort (ACS) | 3 months
  Participation measure:% retained activities.(patient)
Activity Card Sort (ACS) | 6 months
  Participation measure:% retained activities.(patient)
Activity Card Sort (ACS) | 15 months
  Participation measure:% retained activities.(patient)
Six Minutes Walking Test (6MWT) | 3 months
  physical endurance, sub-max test. (patient)
Six Minutes Walking Test (6MWT) | 6 months
  physical endurance, sub-max test. (patient)
Six Minutes Walking Test (6MWT) | 15 months
  physical endurance, sub-max test. (patient)
Health care cost | 3 months
  Evaluation health care cost (patient)
Health care cost | 6 months
  Evaluation health care cost (patient)
Health care cost | 15 months
  Evaluation health care cost (patient)
Checklist Individual Strength subscale fatigue (CIS-fatigue) | 3 months
  Impact of fatigue (patient)
Checklist Individual Strength subscale fatigue (CIS-fatigue) | 6 months
  Impact of fatigue (patient)
Checklist Individual Strength subscale fatigue (CIS-fatigue) | 15 months
  Impact of fatigue (patient)
Health-related Quality of Life: Short Form 36 (SF-36) | 3 months
  Quality of life, used for evaluation of cost effectiveness (patient)
Health-related Quality of Life: Short Form 36 (SF-36) | 6 months
  Quality of life, used for evaluation of cost effectiveness (patient)
Health-related Quality of Life: Short Form 36 (SF-36) | 15 months
  Quality of life, used for evaluation of cost effectiveness (patient)
General Self-Efficacy Scale | 3 months
  Evaluation of the perceived self-efficacy (patient)
General Self-Efficacy Scale | 6 months
  Evaluation of the perceived self-efficacy (patient)
General Self-Efficacy Scale | 15 months
  Evaluation of the perceived self-efficacy (patient)
Hospital Anxiety and Depression Scale (HADS) | 3 months
  Anxiety and depression (patient)
Hospital Anxiety and Depression Scale (HADS) | 6 months
  Anxiety and depression (patient)
Hospital Anxiety and Depression Scale (HADS) | 15 months
  Anxiety and depression (patient)
Zarit Burden Inventory (ZBI) | 3 months
  Perceived caregiver burden (caregiver)
Zarit Burden Inventory (ZBI) | 6 months
  Perceived caregiver burden (caregiver)
Zarit Burden Inventory (ZBI) | 15 months
  Perceived caregiver burden (caregiver)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Cup, dr., Principal Investigator — Radboudumc, department Rehabilitation
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Veenhuizen Y, Satink T, Graff MJ, Geurts AC, Groothuis JT, van Engelen BG, Nijhuis-van der Sanden MW, Cup EH. Mixed methods evaluation of a self-management group programme for patients with neuromuscular disease and chronic fatigue. BMJ Open. 2021 Aug 25;11(8):e048890. doi: 10.1136/bmjopen-2021-048890. PMID 34433601
- [Derived] Veenhuizen Y, Cup EHC, Jonker MA, Voet NBM, van Keulen BJ, Maas DM, Heeren A, Groothuis JT, van Engelen BGM, Geurts ACH. Self-management program improves participation in patients with neuromuscular disease: A randomized controlled trial. Neurology. 2019 Oct 29;93(18):e1720-e1731. doi: 10.1212/WNL.0000000000008393. Epub 2019 Sep 30. PMID 31570565
- [Derived] Veenhuizen Y, Cup EH, Groothuis JT, Hendriks JC, Adang EM, van Engelen BG, Geurts AC. Effectiveness and cost-effectiveness of a self-management group program to improve social participation in patients with neuromuscular disease and chronic fatigue: protocol of the Energetic study. BMC Neurol. 2015 Apr 19;15:58. doi: 10.1186/s12883-015-0314-4. PMID 25913823